CLINICAL TRIAL: NCT06425432
Title: Higher Order Aberration and Relationship With Soft Contact Lens Modulus
Status: Not yet recruiting | Type: Observational
Sponsor: Southern College of Optometry (Other)
Responsible Party: Principal Investigator, Yueren Wang, OD, Assistant Professor, Southern College of Optometry
Other Study IDs: 6733
Record Dates: First submitted 2024-05-15; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Corneal Wavefront Aberration
Keywords: Contact Lens; Higher order aberration; Modulus
MeSH Terms: conditions — Corneal Wavefront Aberration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- CL first: Subject will present wearing habitual contact lenses for the aberrometry measurement. They will then remove their contact lenses and measurement repeated uncorrected.
  Interventions: Device: OVITZ xwave aberrometer
- Glasses first: Subjects will refrain from contact lens wear on day of the visit. Initial aberrometry measurement will be performed uncorrected. They will be then asked to insert their contact lenses and aberrometry measurements repeated.
  Interventions: Device: OVITZ xwave aberrometer

INTERVENTIONS:
Device: OVITZ xwave aberrometer — wavefront aberrometer

SUMMARY:
Higher order aberrations are imperfects in the eye that affect the quality of image projected onto the retina. Soft contact lenses are made of different materials with different stiffness. This study looks to see if the soft contact lens material affects the amount of higher order aberrations in an eye.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Adults > 18 years old regardless of gender, race, or ethnicity
* Habitual single vision soft CL wearer for at least 1 week in any modality.

Exclusion Criteria:

* Multifocal soft CL wear
* GP or ortho K wear in the last 3 months.
* Active eye infections and inflammations.
* Current use of ocular medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults (>18 years old) who are wearing single-vision soft contact lenses will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-20 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in HOA with and without contact lenses | Within the same study visit, measurements will be taken 15 minutes apart to allow for tear film to return to homeostasis after contact lens insertion/removal.
  Measure HOA with contact lenses. And then measure HOA without contact lenses.

SECONDARY OUTCOMES:
Correlation between contact lens modulus and changes in HOA with and without contact lenses | Within the same study visit, measurements will be taken 15 minutes apart to allow for tear film to return to homeostasis after contact lens insertion/removal.
  Evaluate correlation between the lens modulus and changes in HOA

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: 6 months - 3 years after publication
Access Criteria: Upon request

DOCUMENTS (1):
  • Study Protocol (2024-05-13): https://cdn.clinicaltrials.gov/large-docs/32/NCT06425432/Prot_000.pdf